CLINICAL TRIAL: NCT06705881
Title: Efficacy of the Extracorporeal Shock Wave Therapy in Athletes With Patellar Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Abdulhamit Tayfur, physiotherapist/assist prof., Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/1012
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Patellar Tendinopathy; Patellar Tendon Pain
Keywords: exercise; Extracorporeal shock waves therapy; pain; patellar tendinopathy
MeSH Terms: conditions — Motor Activity; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Eccentric exercise program (EEP)
- Intervantion Group (Experimental)
  Interventions: Other: Eccentric exercise program (EEP); Other: ESWT (Extracorporeal Shock Wave Therapy)

INTERVENTIONS:
Other: Eccentric exercise program (EEP) — All participants will perform a 6-week single-leg eccentric squat exercise. It will be performed on an incline board with a 25° incline. It will consist of a single-leg squat, with the downward component (eccentric phase) of the EEP performed using the symptomatic leg and the upward component (concentric phase) using the contralateral leg primarily. If pain occurs during the exercises, athletes will be asked to continue the exercise if they score ≤5 out of 10 on the Visual Acuity Scale (VAS). The exercises will be attempted in the first session of each week, and if no or very little pain is felt, the weight will be increased by 2.5% to increase the intensity of the exercise. Three sets of 15 repetitions per session will be performed twice a day. It will be performed 5 days a week. Participants will be asked to fill out an exercise diary (sets, repetitions, and daily frequency) and return it to the researchers at each follow-up session.
Other: ESWT (Extracorporeal Shock Wave Therapy) — ESWT is a therapy method routinely used in private and public hospitals. Tendinopathy therapy parameters approved by the International Society for Medical Shock Wave Therapy (ISMST) for focused ESWT treatment are: 0.10-0.25 mJ/mm (dosing appropriate to pain), up to a maximum of 5 Hz, 1500-2500 pulses per session, 1-2 weeks apart. Accordingly, in our study, the focused ESWT dosage of the ESWT group will be applied as; 0.10-0.25 mJ/mm (dosing appropriate to pain), 4 Hz, 2000 pulses, 1 session per week for 3 weeks. No exercise will be done on the day of ESWT.
  Arms: Intervantion Group

SUMMARY:
The aim of this study is to investigate the effectiveness of extracorporeal shock wave therapy (ESWT) in addition to eccentric exercise on the clinical outcomes of PT in the treatment of athletes with patellar tendinopathy (PT). Participants will be randomly divided into two groups. The intervention group will receive focus ESWT 3 times a week in addition to 6 weeks of exercise. The control group will be given 6 weeks of exercise. Evaluations will be made at the 3rd and 6th weeks, and at the 3rd, 6th and 12th months. Patient evaluation will begin with obtaining sociodemographic information. Patients' pain level will be assessed using visual analog scale (VAS), tendon pain and function VISA-P, functional capacity; The patients will be assessed with the maximal vertical jump test (MDS), single leg jump distance test (SLHD), single leg squat test (STS) on the incline board, pain catastrophe with the pain catastrophe scale (PCS), kinesiophobia with the Tampa Kinesiophobia Scale (TKS), quality of life short form-12 (SF-12) and physical activity level with the Tegner Activity Scale (TAS).

ELIGIBILITY:
Inclusion Criteria:

* Localized pain in the inferior pole of the patella during single-leg squatting due to load,
* Pain or tenderness with palpation of the patellar tendon,
* Complaints of pain in the patellar tendon due to training, competition or physical activity in the last 6 months,
* Performing sports/physical activities related to jumping and landing,
* Professional and recreational athletes who perform at least 5 and above according to the Tegner Activity score,
* VISA-P scale score <80 out of 100.

Exclusion Criteria:

* Presence of other knee pathologies,
* Known presence of inflammatory joint diseases or familial hypercholesterolemia,
* Daily use of drugs with presumed effects on the patellar tendon (e.g. fluoroquinolones) in the last 12 months,
* Local injection therapy with corticosteroids in the last 12 months,
* Previous patellar tendon rupture,
* Any lower extremity surgery in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Assessment | Baseline
  Age, gender, height, weight, BMI, sports age, occupation, dominant side, affected side, currently doing sports, did they do sports in the past
Visual Analog Scale (VAS) | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  The pain intensity felt by the participants in the knee joint during rest and activity, respectively, will be assessed with VAS. VAS is an easy-to-use scale as it does not have any language and is frequently applied in clinics. Individuals will be asked to describe the pain they feel during the test on a 10 cm scale as "0" (no pain) and "10" (unbearable pain).
VISA-P Questionnaire | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  Assess symptom severity, knee function and sports ability in athletes with PT. VISA-P questionnaire consists of 8 questions. The first 6 questions are to assess symptom severity during sports activities and the last 2 questions ask about sports-related knowledge interaction and participation. The maximum score of the first 7 questions of VISA-P questionnaire is 10 points and the last question is 30 points. Theoretically, the maximum score of VISA-P questionnaire is 100 and the minimum score is 0. The maximum VISA score for an asymptomatic athlete is 100 points.
Maximal vertical jump test | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  The Vertical Jump Test (vertical jump or upright jump) is a commonly performed fitness test to determine an athlete's leg muscle strength or explosive power. The higher the jump, the stronger an athlete's leg muscle/explosive power. The test will be performed with an Optojump.
Single-leg hop distance test (SLHD) | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  The long-distance single-leg hop (SLHD) is the most frequently reported functional test. Participants will be instructed to stand on the leg to be tested, jump as far forward as possible, and land on the same leg. The test procedure will be explained and then demonstrated. Participants will be given a practice run before the main measurement until they become familiar with the test and will be performed three times on both legs, starting with the non-dominant leg. Participants must not have any loss of balance during landing before the jump distance is measured and recorded. Dropping the other foot during the jump or landing, any abnormal movement that causes the supporting leg to move during landing, or touching the ground with the upper extremities will be recorded as a failed attempt. After an unsuccessful attempt, participants will be reminded to maintain balance on the landing leg for two seconds. They will then be allowed to perform a new attempt. The jump test will be considere
Incline board single-leg squat test (EET) | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  The incline board single-leg squat test (EET) is recommended as a provocation test to differentiate patellar tendon pain. The single-leg eccentric squat exercise will be performed on an incline board with a 25° incline (Impellizzeri et al., 2007). The EET will consist of a single-leg squat, with the downward component (eccentric phase) performed with the symptomatic leg and the upward component (concentric phase) primarily using the contralateral leg. The original test was described using a 25° incline board to increase the load on the patellar tendon and avoiding flexion beyond 60°. Localized pain at the inferior pole of the patella is identified as an important diagnostic sign for patellar tendinopathy. Participants will be asked to squat to the point of pain and the squat angles will be measured with a goniometer. Pain levels will be recorded with a VAS. A difference of 2 points on the VAS will be considered the minimal clinically important difference (MCID).

SECONDARY OUTCOMES:
Tegner Activity Scale (TAS) | Baseline
  Tegner activity scale (TAS) is a 1-item instrument that assesses activity levels for sports (competitive or recreational football, basketball, handball, etc.) and occupational activities (light or heavy work). It assesses the patient's work and sports activity level on an 11-level scale, with higher scores representing higher physical activity levels.
Pain Catastrophizing Scale | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  The participants' pain catastrophizing will be assessed using the "Pain Catastrophizing Scale (PCS)". The Turkish version of the "Pain Catastrophizing Scale", which has been reported to reliably predict certain variables such as fear, emotion or thought related to past pain experiences, severe pain, disability and emotional disturbances, will be assessed using the Pain Catastrophizing Scale. The scale consists of 13 questions scored between 0-4 (0=Not at all, 1=Somewhat. 2=Moderately, 3=Severely, 4=Always). An increase in the scale score indicates a high fear of experiencing pain.
Tampa Kinesiophobia Scale | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  TKS is a 17-question checklist and is used in acute and chronic low back pain, fibromyalgia, musculoskeletal injuries, and whiplash-related diseases. The scale uses a 4-point Likert score (1= Strongly disagree, 4= Strongly agree). A total score is calculated after reversing items 4, 8, 12, and 16. The person receives a total score between 17-68. A high score on the scale indicates that the person has high kinesiophobia. The validity and reliability of the questionnaire in Turkish was conducted by Tunca Yılmaz and his colleagues. For chronic pain, a change of 5.6 points is considered clinically significant.
Quality of Life (SF-12) | Baseline, 3 week, 6 week, 3 month, 6 month, 12 month
  SF-12 consists of 8 sub-dimensions and 12 items: physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). While the items related to physical and emotional role are answered as dichotomous (yes or no), the other items have Likert-type options ranging from 3 to 6. The total score of the survey ranges from 0 to 100, with a higher score representing better health.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Breda SJ, Oei EHG, Zwerver J, Visser E, Waarsing E, Krestin GP, de Vos RJ. Effectiveness of progressive tendon-loading exercise therapy in patients with patellar tendinopathy: a randomised clinical trial. Br J Sports Med. 2021 May;55(9):501-509. doi: 10.1136/bjsports-2020-103403. Epub 2020 Nov 20. PMID 33219115